CLINICAL TRIAL: NCT02853149
Title: A Lifestyle Intervention Targeting Enhanced Health and Function for Persons With Chronic SCI in Caregiver/Care-Receiver Relationships: Effects of Caregiver Co-Treatment
Acronym: DRPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, Departments of Neurological Surgery and Physical Medicine & Rehabilitation, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20151065; 90DP0074-01-00 (Other Grant/Funding Number: National Institute on Disability Independent Living, and Rehabilitation Research NIDILRR)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Spinal Cord Injury; Cardiovascular Diseases; Obesity
Keywords: Spinal Cord Injury; disability; obesity; cardiometabolic; Caregiver
MeSH Terms: conditions — Spinal Cord Injuries; Cardiovascular Diseases; Obesity | interventions — Creb3l2 protein, rat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spinal Cord Injury (SCI) (Experimental): Experimental: Lifestyle Intervention This arm will examine whether a twelve month treatment program (one year) for Spinal Cord injury individuals enrolled with their caregivers, can lower body weight, reduce body fat, reduce risk factors for developing heart disease and diabetes, and improve the quality of life using a 6 months of structured lifestyle intervention incorporating education, exercise, diet, and behavioral support.
  Interventions: Behavioral: Spinal Cord Injury (SCI)
- Caregiver Intervention(CCC) (Active Comparator): Lifestyle Intervention This arm will examine whether a twelve month treatment program (one year) enrolled with their Care-receivers( SCI individuals) can lower body weight, reduce body fat, reduce risk factors for developing heart disease and diabetes, and improve the quality of life using a 6 months of structured lifestyle intervention incorporating education, exercise, diet, and behavioral support.
  Interventions: Behavioral: Caregiver Intervention(CCC)
- Caregiver Control (CC) (Placebo Comparator): Placebo: This arm will examine whether a twelve month treatment program (one year) enrolled with their Care-receivers( SCI individuals) can lower body weight, reduce body fat, reduce risk factors for developing heart disease and diabetes, and improve the quality of life. The control group intervention will test benefits of exercise alone while controlling for investigator contact.
  Interventions: Behavioral: Caregiver Control (CC)

INTERVENTIONS:
Behavioral: Spinal Cord Injury (SCI) — The SCI Intervention group will undergo intense exercise, a defined nutrition program, and an educational program taught by the study investigators. The exercise will require them to undergo supervised activity 3 times weekly for 6 months. They will also participate in a series of educational sessions that examine their lifestyle, and modify exercise/nutritional habits. After 6 months they will advance to another 6 months or "extension phase" in which the investigators expect them to continue to exercise up to 3 times per week at our center or at home by using elastic exercise bands (Thera-band) and handles that the Investigators will provide and teach how to use. They will also be expected to continue the modified nutritional program.
  Other Names: Lifestyle program-SCI
  Arms: Spinal Cord Injury (SCI)
Behavioral: Caregiver Intervention(CCC) — The Caregiver Intervention group will undergo intense exercise, a defined nutrition program, and an educational program taught by the study investigators. The exercise will require them to undergo supervised activity 3 times weekly for 6 months. They will also participate in a series of educational sessions that examine their lifestyle, and modify exercise/nutritional habits. After 6 months they will advance to another 6 months or "extension phase" in which the investigators expect them to continue to exercise up to 3 times per week at our center or at home by using elastic exercise bands (Thera-band) and handles that the Investigators will provide and teach how to use. They will also be expected to continue the modified nutritional program.
  Other Names: Lifestyle program-Caregiver Intervention CCC
  Arms: Caregiver Intervention(CCC)
Behavioral: Caregiver Control (CC) — The Caregiver Control group will also discuss ways in which health and fitness can be improved through exercise and nutrition and will also be offered a fully paid membership to the an exercise fitness center to encourage them to exercise and consume a healthy diet. Unlike the Caregiver Intervention group(CCC) the lifestyle recommendations will be provided by internet authorities such as Web Medical(WebMD), the US Department of Agriculture, and the US Department of Human Health Services, which are dependable websites that promote healthy ways of living.
  Other Names: CC
  Arms: Caregiver Control (CC)

SUMMARY:
This study determines in people with chronic SCI the health and functional impact and user acceptance and satisfaction - of a 6-month comprehensive Lifestyle Intervention; the impact and user acceptance/satisfaction of a Complementary Caregiver Curriculum (CCC) on SCI caregiver health and function and whether the complementary caregiver curriculum (CCC) enhances health and functional benefits obtained by the SCI dyadic partner enrolled in the LI program.

DETAILED DESCRIPTION:
The current proposal addresses the compelling problem of cardiometabolic disease risk and functional decline in persons with disability from spinal cord injuries and disease (SCI/D). 'Obesity/overweight' addressed in this project - a major component of cardiometabolic disease risk (CMD) - represents the sole chronic condition whose speed of growth and widespread dispersion parallels pandemics of communicable diseases. Nearly 2/3 of Americans are currently overweight or obese, with a growth rate exceeding 10% in the past decade. The prevalence and impact of obesity is expected to worsen. Obesity-related health risks cross all lines of gender, geographic region, socioeconomic status, race, heritage, and educational level, and are strongly associated with comorbid conditions including: cardiometabolic syndrome, hypertension, diabetes, inflammatory disease, coronary artery disease, congestive heart failure, stroke, osteoarthritis, sleep apnea, depression, cancer, respiratory failure, disorders of coagulation, and degenerative joint disease. All of these disorders are widely reported at elevated prevalence in people with physical disability (PWPD). A study based on pooled data from the 1994-5 National Health Interview Survey, the 1994-5 Disability Supplement, and the 1995 'Healthy People 2000' Supplement reported a 66% higher rate of obesity among PWPD than the general population. A regional study reported that extreme obesity (body mass index [BMI] ≥ 40) was four times more prevalent among PWPD than those without. Prevalence rates for overweight and obesity in persons with chronic SCI/D are equally daunting, and range from 55% to 95.7% of the population. Numerous causes explain accretion of body fat after SCI including sarcopenia leading to loss of metabolically active muscle mass, reduced whole body energy expenditure, restricted choices for exercise conditioning, and a hypercaloric diet. Irrespective of cause, weight gain after disability brings about diminished work capacity, musculoskeletal decline, pain, accelerated cardiovascular diseases (CVD), and progressive life dissatisfaction. Overweight/obesity after SCI/D is also disturbingly co-morbid with dyslipidemia, glucose intolerance, and insulin resistance, a 'pro-inflammatory phenotype, and risks of postprandial lipemia. Increasing body mass (BM) promotes wheelchair injury and dysfunction, imposes significant burdens on self-image and perceived health, and is far more difficult to reverse than obesity occurring in persons without disability. Overweight in particular: a) Poses functional limitations, and restricts physical activity, independence, and community integration; b) affects ease of transferring, joint function, and fracture risk; and, c) compromises 'activities of daily living' (ADLs) in 39% of individuals with SCI. Despite all of these risks and concerns an effective solution to this problem has evaded researchers, clinicians, and stakeholders with SCI.

While an overweight body has implications for health and function of PWPD, it also has an impact on their caregivers. Within the past quarter decade there has been a predictable shift of many health and function related responsibilities to adjuvant providers (i.e., healthcare provider extenders) -- so-called 'caregivers' - who are challenged to administer greater health and functional demands of aging PWPD while they are similarly experiencing health and functional 3 decline accompanying their own aging. This shifting of providers will likely continue, or possibly worsen due to an uncertain future of disability coverage within a tentative American health system. The investigators have already started to observe - yet not fully comprehend - the many complex difficulties imposed by aging on PWPD and their caregivers, and speculate how to effectively intervene on them. Unlike caregivers for persons with Alzheimer's disease and Parkinson's disease, caregivers of people with wheelchair dependency are required to be more physically active, lift/push/roll an impaired body far more often, and often assume caregiving responsibilities earlier in the life of PWPD. While clinicians and researchers often focus on the person with disability, their caregiver can be left out of the care plan. It is thus not surprising that pain, anxiety, and depression among caregivers of PWPD is exceedingly prevalent.

Encouraging evidence already suggests an important role for primary and secondary lifestyle intervention (LI) in the form of weight-lessening and fitness-promoting nutrition and exercise to improve health and function of people aging with disability. Comprehensive LI programs of exercise, nutrition, and behavioral support for people without disabilities have been designed and systematically tested in multi-center clinical trials, and have been found effective in the short term for promoting weight loss and lessening conversion rates to frank diabetes. The LI programs have been compared against pharmacotherapy and have actually been found more effective. Programmatic modifications made for community deployment of the LI plans, and testing of long-term follow-up have shown remarkable success in sustaining - or even further improving - benefits obtained during initial treatment. These research findings make LI programs of weight-loss promoting reconditioning exercise, nutrition, and behavioral support legitimate candidates for testing in PWPD, although no studies have ever done so. Moreover, the impact of these interventions on caregiver burden has never been examined, although it is reasonable to conjecture that loss of body BM and improved fitness/function of care-receivers would reduce global caregiver burden. Further, evidence supports lifestyle and health benefits to the care-receiver when a caregiver is enrolled in a linked behavioral intervention program, making the relationship of the dyadic partners in benefiting one another through coordinated intervention an intriguing intervention benefit.

To: a) address the concerning problem of overweight/obesity after SCI, b) better understand its impact on health and function of persons with SCI and their caregivers, and c) intervene on these hazards where inaction would forecast additional decline, the investigators will conduct a randomized, controlled, multi-center intervention study examining persons with disability from SCI and their caregivers, who will together be enrolled as dyadic partners. Key questions will address whether: a) people with disability from SCI benefit from the LI plan through improved health and function, b) caregivers of people with disability from SCI benefit from the LI plan through their own improved health and function, c) co-participation of a caregiver partner in a LI curriculum provides a cross benefit for their partner, and d) benefits of clinical intervention are long-lasting with minimal supervision. The investigators will use an intervention for all participants with SCI that is modeled after the Diabetes Prevention Program (DPP) that incorporates population-appropriate exercise, nutrition, and behavioral support. Caregivers (linked with their partners) will be randomized to either 'behavioral support' or a 'control condition'. Clinical training will take place for 6 months and then be followed by a 6-month minimally supervised extension phase. Outcomes tested for participants with SCI will focus on domains of health and function reflected by fitness, cardioendocrine risk and inflammatory stress; multi-dimensional function and pain; Sol and independence; and self-efficacy, program acceptance, and life satisfaction. Outcomes tested for caregivers will focus on multidimensional function and pain; and, Quality of Life (QoL) and independence, the latter including perceived caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

a. Inclusion Criteria:

1. Men and Women with SCI/D > 1 year, aged 18-70 years.
2. American Spinal Injury Association (AIS) Impairment scale A-D Spinal Cord Levels C5-L1
3. Any one or more of the following:

   1. Waist circumference >94 cm (37 inches)
   2. BMI ≥ 21 kg/m2
   3. Fasting dyslipidemia (either; High-density lipoprotein cholesterol (HDL-C)≤ 40mg/dL (men)/≤50 mg/dL (women), or Triglycerides (TG) ≥ 150 mg/dL).

      AND,
   4. Linked with caregivers: Men and women 18-70 years who consent to co-enroll in the study with their partner. Caregivers are defined as: Family member, significant others or friends living with a disabled (SCI/D) partner who provide social and/or physical support including personal assistance, routine emotional encouragement and/or social interaction.

Exclusion Criteria:

* Exclusion Criteria for Participants with SCI/D:

  1. Participating in at least 30 minutes of moderate intensity physical activity on at least three days of the week for at least three months.
  2. Diet involving moderate caloric restriction for at least 6 months resulting in weight loss/gain ≥ 10% of total body mass
  3. Surgery within 3 months.
  4. Grade 3-4 pressure ulcer within 3 months;
  5. limb pain that limits exercise
  6. recurrent acute infection or illness
  7. pregnancy
  8. previous myocardial infarction (MI), or cardiac surgery
* Exclusion Criteria for Caregiver Participants:

  1. Participating in at least 30 minutes of moderate intensity physical activity on at least three days of the week for at least three months
  2. Diet involving moderate caloric restriction for at least 6 months.
  3. weight loss/gain of 10% within the preceding 6 months
  4. Surgery within 3 months.
  5. upper limb pain that limits exercise
  6. pregnancy
  7. Previous myocardial infarction (MI), cerebrovascular accident (CVA) or cardiac surgery that limits exercise.
  8. Type I or II diabetes by World Health Organization (WHO) criteria
* Other exclusions applying to groups:

  1. The following drugs: anti-hyperglycemic agents, and lipid-altering agents within the past 6 months. Women who become pregnant will be advised to notify study personnel, will be tested, and if found to be pregnant discharged from the trial. There is no harm caused by exercise and diet in early pregnancy. Women must wait 6 months after child delivery to enter the study - a criterion of the Diabetes Prevention Program.
  2. Individuals with a diagnosis of pre-diabetes if, after 2 months of intervention the following diagnostic criteria of the American Diabetes Association criteria (ADA) are observed:

Fasting Blood Glucose (FBG) 110-126mg/dL after a fast of 8 hours OR 2 hyperglycemia symptoms (i.e. Polyuria, polydipsia and unexplained weight loss) and a causal plasma glucose ≥200 mg/dL. In the absence of unequivocal hyperglycemia, these criteria will be confirmed by repeat testing per (ADA) criteria. Should repeat testing confirm diabetes, subjects will be discharged and referred for medical treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06-26 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Fitness indicators as measured by Body Mass index (BMI)- | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months.
  Body Mass index will be calculated with the respective formula after collecting Height (supine position) and weight (calibrated scale), expressed in kg/m2

SECONDARY OUTCOMES:
Change from baseline in Cardioendocrine and Global Cardiovascular risk by surrogate blood measures of the Homeostasis Model Assessment -Insulin Resistance (HOMA 2-IR) in SCI individuals and caregivers (unitless) | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results obtained from wash in ( -2 months) and baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.
Change from baseline in Cardioendocrine and Global Cardiovascular risk by surrogate blood measures of the Total Cholesterol(TC): High Density high-density lipoprotein(HDL) ratio in SCI individuals and caregivers | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results obtained from wash in ( -2 months) and baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.
Change in Inflammatory state cytokines by surrogate blood measures in SCI and Caregivers of Interleukin 6 (IL-6) and Interleukin (IL-1) tests | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results obtained from wash in ( -2 months) and baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.
Change in Inflammatory state cytokines by surrogate blood measures in SCI and Caregivers of Tumor necrosis factor alpha (TNF-α) | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results obtained from wash in ( -2 months) and baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.
Change from baseline in Fitness indicators as measured by Endurance-maximal oxygen consumption (Vo2 peak test)individuals and their caregivers | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results obtained from wash in ( -2 months) and baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.
Change from baseline in Fitness indicators as measured by Strength- one-repetition maximum test ( 1RM) in SCI individuals and their caregivers | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results obtained from wash in ( -2 months) and baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.

OTHER OUTCOMES:
Change from baseline in Multi-dimensional Pain-The West Haven-Yale Multi-dimensional Pain Inventory (MPI-SCI) | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results scores obtained from wash in ( -2 months) and baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.
Change from baseline in Caregiver Function- Patient-Reported Outcomes Measurement Information System (PROMIS) | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results scores obtained from wash in ( -2 months) and baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.
Change from baseline in Basic Pain and Classification after SCI -The International SCI Basic Pain Data Set (ISCIBPDS) | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results scores obtained from baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.
Change from baseline in Neuropathic pain as measured by The Neuropathic Pain Symptom Inventory (NPSI) | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results scores obtained from baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.
Change from baseline in Multi-dimensional Pain-The West Haven-Yale Multi-dimensional Pain Inventory (MPI) | -2 Months (Wash) to Baseline (0 Months); to 6 Months and 12 Months and Baseline (0 months) to 6 Months and 12 Months
  Change will be calculated using the difference in results scores obtained from baseline ( 0 months) vs. each period of testing (6 and 12 months) and it will be expressed in percentage % of change over that period.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Craig Hospital, Englewood, Colorado
  - University of Miami- The Miami Project to Cure Paralysis, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bigford GE, Lehmann DA, Betancourt LF, Maher JL, Mendez AJ, Nash MS. Modification of the Diabetes Prevention Program Lifestyle Intervention in Persons with Spinal Cord Injury: Efficacy for Reducing Major Cardiometabolic Risks, Increased Fitness, and Improved Health-Related Quality of Life. J Spine Res Surg. 2024;6(1):10.26502/fjsrs0070. doi: 10.26502/fjsrs0070. PMID 39309246
- [Derived] Bigford GE, Lehmann DA, Mendez AJ, Nash MS. The Impact of Caregiver/Care-Receiver Co-Treatment in a Therapeutic Lifestyle Intervention for Chronic Spinal Cord Injury: A Comparative Case Series. Ann Case Rep. 2024;9(2):10.29011/2574-7754.101755. doi: 10.29011/2574-7754.101755. PMID 39308936
- [Derived] Bigford GE, Betancourt LF, Charlifue S, Nash MS. Therapeutic Lifestyle Intervention Targeting Enhanced Cardiometabolic Health and Function for Persons with Chronic Spinal Cord Injury in Caregiver/Care-Receiver Co-Treatment: A Study Protocol of a Multisite Randomized Controlled Trial. Int J Environ Res Public Health. 2023 Sep 25;20(19):6819. doi: 10.3390/ijerph20196819. PMID 37835090